CLINICAL TRIAL: NCT02443558
Title: Brainwave Control of a Wearable Robotic Arm for Rehabilitation and Neurophysiological Study in Cervical Spine Injury
Acronym: CSI:Brainwave
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Cervical Spine Research Society (Other)
Responsible Party: Principal Investigator, Panos Bamidis, Assistant Professor, Aristotle University Of Thessaloniki
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 90886
Record Dates: First submitted 2015-05-05; First posted 2015-05-14 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Spinal Cord Injuries
Keywords: Robotics; Cerebral cortex; Brain waves; Electroencephalography; Rehabilitation; Brain-Computer Interfaces
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Complete Injury (Experimental): Patients suffering from complete injury at the cervical spinal cord level (ASIA Impairment Scale A).
  Brain-Computer Interface control of robotic arms. MERCURY v2.0 robotic arms.
  Interventions: Other: Brain-Computer Interface control of robotic arms.; Device: MERCURY v2.0 robotic arms
- Incomplete Injury (Experimental): Patients suffering from incomplete injury at the cervical spinal cord level (ASIA Impairment Scale B,C,D,E).
  Brain-Computer Interface control of robotic arms. MERCURY v2.0 robotic arms
  Interventions: Other: Brain-Computer Interface control of robotic arms.; Device: MERCURY v2.0 robotic arms
- Non-cervical injury (Active Comparator): Patients suffering from complete or incomplete injury of the spinal cord at a level other than the cervical (thoracic or lumbar).
  Brain-Computer Interface control of robotic arms. MERCURY v2.0 robotic arms
  Interventions: Other: Brain-Computer Interface control of robotic arms.; Device: MERCURY v2.0 robotic arms
- Healthy participants (Active Comparator): Healthy participants, age and sex matched to those of the other Arms.
  Brain-Computer Interface control of robotic arms. MERCURY v2.0 robotic arms
  Interventions: Other: Brain-Computer Interface control of robotic arms.; Device: MERCURY v2.0 robotic arms

INTERVENTIONS:
Other: Brain-Computer Interface control of robotic arms. — The patients will be trained to modulate self-paced Visual Motor Imagery (VMI) and Kinesthetic Motor Imagery (KMI) under EEG recording in order to achieve BCI-control of a custom-built bimanual arms robot (MERCURY v2.0). In KMI they will be asked to modulate brain waves in order to learn to control the BCI and in VMI they will additionally be projected a visual cue (representation of the intended movement).
Device: MERCURY v2.0 robotic arms — MERCURY v2.0 robotic arms is a non-commercial 6-degree-of-freedom anthropomorphic bimanual robotic arms device that was built and developed by the research team of the Medical Physics Lab.
  Other Names: robotic arms

SUMMARY:
CSI:Brainwave is a multidisciplinary neurophysiological project, developed by the Lab of Medical Physics, School of Medicine, Aristotle University of Thessaloniki and supported by two Neurosurgical Departments. The project officially commenced on April 2014 and the first year was awarded the 2013 Mario Boni Research Grant by the Cervical Spine Research Society-European Section (CSRS-ES). The website for the project can be accessed at http://medphys.med.auth.gr/content/csi-brainwave.

The investigation's primary objectives include the development, testing and optimization of a mountable robotic arm controlled with wireless Brain-Computer Interface, the development and validation of a self-paced neuro-rehabilitation protocol for patients with Cervical Spinal Cord Injury and the study of cortical activity in acute and chronic spinal cord injury.

DETAILED DESCRIPTION:
CSI:Brainwave project's full title is <Brainwave control of a wearable robotic arm for rehabilitation and neurophysiological study in Cervical Spine Injury> . It is a multidisciplinary neurophysiological project, developed by the Lab of Medical Physics and supported by two Neurosurgical Departments.

The CSI:Brainwave project involves:

1. A clinical study for rehabilitation of patients with Cervical Spinal Cord Injury (CSCI), using a Brain-Computer Interface (BCI) controlled robotic arms device.
2. A secondary off-line neurophysiological analysis of cortical activation, connectivity and plasticity in patients with CSCI undergoing motor imagery (MI) practice.

Milestones of the study:

1. The investigators aim to develop, test and optimize a mountable robotic arm controlled with wireless BCI.
2. The investigators aim to develop and validate self-paced neuro-rehabilitation protocols for patients with CSCI.
3. The investigators aim to identify and study the neurophysiological functionality and alteration of cortical activity in acute and chronic CSCI.

The CSI: Brainwave project aims at allowing patients suffering from tetraplegia due to CSCI to perform brainwave modulation, practicing Kinesthetic Motor Imagery (KMI) and Visual Motor Imagery (VMI), as well as offering neurofeedback with the form of control of a 6-degree-of-freedom, anthropomorphic bimanual robotic arms device. The project aims at demonstrating the added value of neurofeedback for rehabilitation and/or motor restoration of CSCI patients and allow for elaborate recordings of motor-related brain activity during motor tasks of the upper and lower extremities.

The robotic arms are designed to mount on a frame that acts as a docking space for the participants' armchair/wheelchair and will be directly controlled by the participants using a BCI module. The investigators aim to further modify the robotic device in order to render it mountable on the participants' actual arms.

The largest portion of the first project year was devoted to the development of robotics and the Brain-Computer Interface module of the study. The MERCURY v2.0 robotic arms is a non-commercial 6-degree-of-freedom anthropomorphic bimanual robotic arms device that was built and developed by the research team of the Medical Physics Lab. The robot was further engineered to accommodate the needs of the CSI:Brainwave project. The investigators aim to use the Emotiv EPOC wireless EEG headset and software for the development and control of the BCI module in this study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Spinal Cord Injury (SCI evaluated by ASIA Impairment Scale).
* Healthy participants (age and gender matched to SCI patients)
* Sufficient documentation of the injury in case of patients (neurological examination, MRI scan of the injury level, optional additional CT or x-rays).
* Signed informed consent (patients and healthy individuals).

Exclusion Criteria:

* Other neurological condition that has a possibility to significantly affect the neurological status of the participants (or) the ability to control a BCI (or) the neurophysiological recordings:

  * Traumatic brain injury
  * Central Nervous System tumors
  * Multiple Sclerosis
  * Amyotrophic Lateral Sclerosis
  * Parkinson's disease
  * Refractory Epilepsy
* Participation during the last 3months in an another interventional study, the effects of which could affect this study's observations.
* Other grave medical condition that could affect the participation (or) the safety of the participants:

  * Cardiac deficiency
  * Pulmonary deficiency
* Hearing and visual impairments that can affect the participant's understanding of the intervention and performance.
* Illegal drug use
* Chronic alcoholism

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
BCI control (yes/no). (ability of participants to modulate brainwave activity in order to achieve control of the BCI) | 1 month after first participation in a BCI session.
  The ability of participants to modulate brainwave activity in order to achieve control of the BCI.
  BCI control is evaluated as achieved or not (there are cases of BCI-illiteracy when the participants cannot modulate their brainwaves in order to control the BCI).

SECONDARY OUTCOMES:
Initial Functional Improvement (Greek translation of the Spinal Cord Independence Measure, version III (g-SCIM-III) | 6 months after first participation in a BCI session.
  Daily functionality as measured by the Greek translation of the Spinal Cord Independence Measure, version III (g-SCIM-III).
Long-term Functional Improvement (Greek translation of the Spinal Cord Independence Measure, version III (g-SCIM-III) | 1 year after first participation in a BCI session.
  Daily functionality as measured by the Greek translation of the Spinal Cord Independence Measure, version III (g-SCIM-III).
BCI performance (classification accuracy (percentage of voluntary non-erroneous commands to overall number of detected commands) and by bit rate (number of commands per minute) | 6 months after first participation in a BCI session.
  Achieved performance on BCI at conclusion of BCI sessions for each participant. Measured by classification accuracy (percentage of voluntary non-erroneous commands to overall number of detected commands) and by bit rate (number of commands per minute).

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Bamidis, PhD, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- Lab of Medical Physics, Faculty of Medicine, Aristolte University of Thessaloniki, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Athanasiou A, Klados MA, Pandria N, Foroglou N, Kavazidi KR, Polyzoidis K, Bamidis PD. A Systematic Review of Investigations into Functional Brain Connectivity Following Spinal Cord Injury. Front Hum Neurosci. 2017 Oct 25;11:517. doi: 10.3389/fnhum.2017.00517. eCollection 2017. PMID 29163098
- [Background] Athanasiou A, Klados MA, Styliadis C, Foroglou N, Polyzoidis K, Bamidis PD. Investigating the Role of Alpha and Beta Rhythms in Functional Motor Networks. Neuroscience. 2018 May 15;378:54-70. doi: 10.1016/j.neuroscience.2016.05.044. Epub 2016 May 27. PMID 27241945
- [Result] Athanasiou A, Xygonakis I, Pandria N, Kartsidis P, Arfaras G, Kavazidi KR, Foroglou N, Astaras A, Bamidis PD. Towards Rehabilitation Robotics: Off-the-Shelf BCI Control of Anthropomorphic Robotic Arms. Biomed Res Int. 2017;2017:5708937. doi: 10.1155/2017/5708937. Epub 2017 Aug 29. PMID 28948168
- [Result] Athanasiou A, Arfaras G, Pandria N, Xygonakis I, Foroglou N, Astaras A, Bamidis PD. Wireless brain-robot interface: user perception and performance assessment of spinal cord injury patients. Wireless Communication and Mobile Computing, 2017: 2986423, 2017 https://doi.org/10.1155/2017/2986423
- [Derived] Athanasiou A, Terzopoulos N, Pandria N, Xygonakis I, Foroglou N, Polyzoidis K, Bamidis PD. Functional Brain Connectivity during Multiple Motor Imagery Tasks in Spinal Cord Injury. Neural Plast. 2018 May 2;2018:9354207. doi: 10.1155/2018/9354207. eCollection 2018. PMID 29853852